CLINICAL TRIAL: NCT07186114
Title: A Prospective Study on the Therapeutic Outcomes of Mebo and Tantum Verde in Patients With Oral Mucositis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Adel Azab, Lecturer of Oral Medicine and Periodontology- Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MeboOM
Record Dates: First submitted 2025-09-05; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Oral Mucositis (Ulcerative) Due to Radiation
Keywords: Moist exposed burn ointment; Oral Mucositis Assessment Scale
MeSH Terms: conditions — Stomatitis; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEBO (Experimental)
  Interventions: Drug: MEBO Wound Ointment (MEBO)
- Tantum Verde (Active Comparator)
  Interventions: Drug: Tantum Verde® mouthwash

INTERVENTIONS:
Drug: MEBO Wound Ointment (MEBO) — MEBO® 0.25% Ointment (Gulf Pharmaceutical Industries) to be applied four times a day for two weeks
  Arms: MEBO
Drug: Tantum Verde® mouthwash — Tantum verde (EIPICO®) mouthwash. Patients were asked to swish it for at least five minutes, four times daily for two weeks.
  Arms: Tantum Verde

SUMMARY:
This study aimed to assess the efficacy of MEBO® in the treatment of already established oral mucositis. This is a randomized controlled clinical trial. The study included 36 patients with established oral mucositis, divided into two groups. Patients were randomly allocated to either receive topically applied MEBO® ointment or Benzydamine Hydrochloride (Tantum Verde) mouthwash three times a day for two weeks. We assessed the World Health Organization mucositis score (WHO), the Oral Mucositis Assessment Scale (OMAS), and the Patient-Reported Oral Mucositis Symptom (PROMS) score at baseline, and after one and two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who later on during radiotherapy developed oral mucositis with a severity of WHO score II or more and were over 18 years were then included in the study and allocated to one of the treatment groups .

Exclusion Criteria:

* We excluded patients who were receiving any prophylactic agents and/or corticosteroids and those who would not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2024-12-14 (Actual)

PRIMARY OUTCOMES:
WHO oral mucositis score | We assessed patients for the three outcomes at baseline, one week and at the end of the study period which is two weeks
  The WHO oral mucositis score is an ordinal scale. The grades are as follows: Grade 0 is no mucositis, Grade 1 is soreness and/or erythema, Grade 2 involves ulcers and the ability to eat solids, Grade 3 indicates ulcers and the need for a liquid diet, and Grade 4 signifies ulcers with no possible oral alimentation

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Dentistry - Cairo University, Cairo
  - Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT07186114/Prot_SAP_ICF_000.pdf